CLINICAL TRIAL: NCT03135483
Title: Assessment of Acute Kidney Injury as a Risk Factor for Myocardial Injury After Non Cardiac Surgery in Critical Patients
Acronym: clinical audit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Safwat, assiut, Assiut University
Other Study IDs: Assiut university1711
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Assesse Prevalence of Acute Kidney Injury and Myocardial Injury After Non Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) affects approximately 20% of hospitalized patients and up to 67% of those admitted to an intensive care unit (ICU), making it among the most common organ dysfunctions among the critically ill.Major adverse cardiac events (MACE) after non cardiac surgery are a leading cause of morbidity and mortality. The reported incidence of postoperative myocardial infarction (POMI) among patients undergoing noncardiac surgery is between 3% and 6%.The aim of this study is to Identify the impact of acute kidney injury on the development of myocardial injury after non cardiac surgery and to correlate it with other risk factors of for MINS.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is classically described as an abrupt or rapidly reversible reduction in the excretion of nitrogenous waste products, including urea, nitrogen, and creatinine. Acute kidney injury (AKI) affects approximately 20% of hospitalized patients and up to 67% of those admitted to an intensive care unit (ICU), making it among the most common organ dysfunctions among the critically ill. Depending on severity, AKI contributes to short-term mortality rates between 40% and 70%, and survivors are at increased risk for chronic kidney disease. Because surgical care and perioperative events and comorbidities interact to contribute to renal dysfunction in different patterns than in nonsurgical patients, surgical patients have unique risk factors for renal dysfunction.

Major adverse cardiac events (MACE) after non cardiac surgery are a leading cause of morbidity and mortality. The reported incidence of postoperative myocardial infarction (POMI) among patients undergoing noncardiac surgery is between 3% and 6%. Early recognition and timely treatment of POMI after surgery are very important. Therefore, routinemonitoring of cardiac troponin has been recommended to identify patients at risk of early postoperative cardiovascular events after surgery. Myocardial injury after noncardiac surgery (MINS) is defined as follows: myocardial injury caused by ischemia (that may or may not result in necrosis), has prognostic relevance, and occurs duringor within 30 days after noncardiac surgery. MINS can be measured by postoperative troponin elevation in the presence or absence of clinical symptoms. MINS occurs in 8% to 22% of adults undergoing major non cardiacsurgery. To date, there have been few studies investigatingthe risk factors of MINS in critical patients.

The postoperative AKI is a new risk factor of MINS in critical patients, and the impact of AKI on MINS has not been evaluated in previous studies.

It is unclear by what mechanisms AKI influences theMINS in critical patients. A possible explanation of this finding is that in patientswith postoperativeAKI, disturbed autonomic nerve functions may induce postoperative hypotension and hypoperfusion, which may lead to MINS .

Other idependent risk factors for myocardial injury after non cardiac surgery such as emergency surgery and long time operation.The aim of this study is to Identify the impact of acute kidney injury on the development of myocardial injury after non cardiac surgery and to correlate it with other risk factors of for MINS.

ELIGIBILITY:
Inclusion Criteria:

* -All patients aged 18 years or more undergoing non cardiac surgery under general or spinal anesthesia and expected length of postoperative hospital stay of at least 48 hour.

Exclusion Criteria:

* -Pregnancy
* Perioperative myocardial injury caused by a documented nonischemic etiology (eg, pulmonary embolism, sepsis, cardio version),
* Heart failure NYHA class III and IV.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult above 18 years undergoe non cardiac surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Acute Kidney Injury as a Risk Factor for Myocardial Injury after non Cardiac Surgery in Critical Patients | one year
  assessment of a risk factor

IPD SHARING:
Plan to Share IPD: Undecided
adult above 18years admitted to assiut university hospital intensive care units after non cardiac surgery